CLINICAL TRIAL: NCT00210587
Title: A Pilot Study to Evaluate the Response Rate of Epoetin Alfa (PROCRIT) at 80,000 Units Every Three Weeks in Anemic Patients With Cancer Not Receiving Chemotherapy or Radiation Therapy
Brief Title: An Efficacy and Safety Study for Epoetin Alfa (PROCRIT) in Cancer Patients Not Receiving Chemotherapy or Radiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003223
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-05

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; Neoplasms; hemoglobin level
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of epoetin alfa (PROCRITÂ®) administered 80,000 Units every three weeks in cancer patients that are not receiving chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
The current approved dosage for epoetin alfa is 40,000 Units once per week with an escalation to 60,000 Units once per week if the response is inadequate after four weeks of treatment at 40,000 Units. This dosing scheme, while proven to be efficacious, is often inconvenient for both patients and medical personnel. This is an open-label, non-randomized, multi-center pilot study with the objective to investigate the efficacy of epoetin alfa (PROCRIT®) with regard to hematopoietic response when administered at 80,000 Units subcutaneously every three weeks in anemic patients with cancer not receiving chemotherapy or radiation therapy. Patients will receive two epoetin alfa injections (40,000 Units per injection) under the skin once every three weeks for a maximum of 13 weeks, totalling a maximum of four treatments. Doses may be reduced depending on the patients' hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin value of <= 11 g/dL unrelated to transfusion
* Patients must not be receiving or planning to receive chemotherapy or radiotherapy within the 13-week study period. However, patients receiving hormonal therapy or non-myelosuppressive therapies are allowable
* Female patients with reproductive potential must have a negative serum pregnancy test at screening
* Patients must have signed an informed consent

Exclusion Criteria:

* Uncontrolled hypertension
* History (within 6 months) of uncontrolled cardiac arrhythmias, or history of pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic coagulation disorder
* Transfusion within 28 days prior to first dose
* Planned chemotherapy or radiation during study and no prior chemotherapy within 8 weeks or radiation within 4 weeks of study entry
* No prior treatment with Epoetin alfa or any other erythropoietic agent within the previous two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-02; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients that achieved a hematopoietic response, defined as a Hb increase >= 2 g/dL and/or Hb = 12 g/dL during the study independent of transfusion within 28 days

SECONDARY OUTCOMES:
Transfusion requirements, change in Quality of Life scores measured by LASA & FACT-An, mean time to hematopoietic response (defined in Primary Endpoint) & mean time to >= 1g/dL change in Hb from baseline. Incidence of adverse events for study duration

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Pilot Study to Evaluate the Response Rate of PROCRIT (epoetin alfa) at 80,000 Units Every Three Weeks in Anemic Patients with Cancer Not Receiving Chemotherapy or Radiation Therapy. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=512&filename=CR003223_CSR.pdf